CLINICAL TRIAL: NCT00749476
Title: Reformulated BeneFIX Efficacy and Safety After Conversion From a pdFIX
Brief Title: Study Evaluating BeneFIX in Patients With Haemophilia B, Previously Treated With Plasma Derived Factor IX
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Responsible Party: Wyeth (Registry Contact: Clinical Trial Registry Specialist), Wyeth
Allocation: Non-Randomized | Model: Single Group | Masking: None
Other Study IDs: 3090X1-4405
Record Dates: First submitted 2008-09-08; First posted 2008-09-09 (Estimated); Results first posted 2010-06-29 (Estimated); Last update posted 2011-06-08 (Estimated); Status verified 2011-06

CONDITIONS: Hemophilia B
MeSH Terms: conditions — Hemophilia B

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental)
  Interventions: Biological: Factor IX recovery

INTERVENTIONS:
Biological: Factor IX recovery

SUMMARY:
The purpose of this study is to collect data around the period of the conversion from plasma-derived Factor IX (pdFIX) to BeneFIX. The main information collected will be: a retrospective history of the bleedings in the 3-month period before the conversion, the recovery with pdFIX just before the conversion and with BeneFIX just after the conversion, and a prospective history of the bleedings in the 3 month period following the conversion.

DETAILED DESCRIPTION:
The switch to BeneFIX has already been decided by the investigator. Patients will be followed up to 3 months after the switch.

ELIGIBILITY:
Inclusion Criteria:

* Moderately to severe haemophilia B patient (FIX activity < or equal to 2%) for whom the switch from pdFIX to BeneFIX has already been decided by the investigator
* Previously treated patients (PTP) with > or equal to 150 ED to any FIX product
* Male patients, aged > or equal to 12 years
* Absolute CD4 count > or equal to 300/microL
* Normal platelet count (> or equal to 100 000/microL)
* Patient is in a non-bleeding state and has not received any coagulation FIX within five (5) days of recovery
* Written informed consent obtained prior to study entry (for patients aged < 18 years, parents' signature or subject legally acceptable representative obtained prior to study entry)

Exclusion Criteria

* Any other known bleeding disorder in addition to haemophilia B
* History of, or current detectable factor IX inhibitor (> or equal to 0.6 BU by Bethesda inhibitor assay)
* History of anaphylaxis to any coagulation factor IX
* Patient with a known hypersensitivity to hamster protein
* Patient with a hypersensitivity to the active substance or to any of the excipients
* Patient unable to be off FIX replacement therapy for at least 5 days without bleeding Patient with hepatic or renal impairment (ALT [SGPT] and AST [SGOT] > 5 x Upper Limit Normal (ULN), total bilirubin > 20mg/l, albumin < 25 g/l, prothrombin time > 1.25 x ULN, serum creatinine > 1.25 x ULN)
* Treatment with any investigational drug or device within the past 30 days
* Any condition that, in the Investigator's judgment, makes participation in the study not advisable

Min Age: 12 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2008-04; Primary Completion 2009-01 (Actual); Study Completion 2009-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Wyeth is now a wholly owned subsidiary of Pfizer
Locations (8):
- France (8):
  - Dr. Lambert, Le Kremlin-Bicêtre
  - Pr Chambost, Marseille
  - Dr. Hassoun, Montmorency
  - Pr Schved, Montpellier
  - Dr. Rothschild, Paris
  - Dr. Duillet, Rennes
  - Dr. Borg, Rouen
  - Pr Gruel, Tours

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were recruited in France from May 2008 to January 2009.
Pre-assignment Details: Before enrollment there was up to a 14 day screening period and the investigator reviewed the subject's medical history and medications to ensure that the subject was in good health and met all of the inclusion criteria and none of the exclusion criteria.
Groups:
- BeneFIX: Plasma-derived FIX recovery with a dose of 50 ± 5 IU/kg before the conversion, BeneFIX recovery with a dose of 50 ± 5 IU/kg after the conversion, treatment with BeneFIX during the next 3 months.
Period: Overall Study
Arm/Group | BeneFIX
Started | 1
Completed | 1
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | BeneFIX
Number analyzed (Participants) | 1
Age Continuous [Mean (Standard Deviation); unit: years] | 27.0 (0.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Reporting Efficacy
Description: Clinical efficacy was measured by number/location of bleeding episodes, number of injections per bleeding, factor IX consumption, global assessment of efficacy by investigator and patient; biological efficacy (recovery) with BeneFIX was measured just after conversion.
Time Frame: 4 months
Population: Intent to Treat (ITT) population. Due to low number of subjects that completed, no descriptive statistics for the efficacy endpoints are provided.
Measure: Number; unit: Participants
Arm/Group | BeneFIX
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Arm/Group | BeneFIX
Serious Adverse Events (participants affected / at risk) | 1/1
Other Adverse Events (participants affected / at risk) | 1/1
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | BeneFIX (N=1)
Herpes simplex type-2 (HSV-2) meningitis (Infections and infestations) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | BeneFIX (N=1)
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 1
Diarrhea (Gastrointestinal disorders) | 1
Acute renal failure (Renal and urinary disorders) | 1
Lower back pain (Musculoskeletal and connective tissue disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The PIs agreed to allow the sponsor 60 days to review and require changes to presentations or publications but only to protect confidential information and intellectual property, and for the sponsor to file a patent application, as applicable. The PIs also agreed for data to be presented first as a joint, multi-center publication.